CLINICAL TRIAL: NCT05610124
Title: Postprandial Glycemia and Satiety of Meals With Potatoes, With and Without Protein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 43406
Record Dates: First submitted 2022-10-24; First posted 2022-11-09 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Glycemic Control; Satiety Response; Appetite Regulation; Diabetes; Obesity
Keywords: Glycemic Control; Satiety; Appetite; Potato; Protein quality; Blood glucose; Insulin; Ghrelin; Nutrition
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Study Design:
  The experiment follows a randomized, cross-over, repeated measures acute trial design.
Who Masked: Participant
Masking Description: True double blinding is not feasible in these study designs. Inherent differences in taste, smell, look and preparation of the various treatments are conspicuous and thus not possible to double-blind. This study is an ad libitum study to simulate a mealtime at home.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Ad libitum full-fat French fries with beef meatballs (Experimental): Ad libitum carbohydrate side with fixed amount of protein: Ad libitum full-fat French fries with beef meatballs (25 g protein)
  Interventions: Other: Ad libitum full-fat French fries with beef meatballs
- Ad libitum instant mashed potatoes with beef meatballs (Experimental): Ad libitum carbohydrate side with fixed amount of protein: Ad libitum instant mashed potatoes with beef meatballs (25 g protein)
  Interventions: Other: Ad libitum instant mashed potatoes with beef meatballs
- Ad libitum macaroni pasta with beef meatballs (Experimental): Ad libitum carbohydrate side with fixed amount of protein: Ad libitum macaroni pasta with beef meatballs (25 g protein)
  Interventions: Other: Ad libitum macaroni pasta with beef meatballs
- Ad libitum full-fat French fries with vegetarian substitute meatballs (Experimental): Ad libitum carbohydrate side with fixed amount of protein: Ad libitum full-fat French fries with vegetarian substitute meatballs (25 g protein)
  Interventions: Other: Ad libitum full-fat French fries with vegetarian substitute meatballs
- Ad libitum instant mashed potatoes with vegetarian substitute meatballs (Experimental): Ad libitum carbohydrate side with fixed amount of protein: Ad libitum instant mashed potatoes with vegetarian substitute meatballs (25 g protein)
  Interventions: Other: Ad libitum instant mashed potatoes with vegetarian substitute meatballs
- Ad libitum macaroni pasta with vegetarian substitute meatballs (Experimental): Ad libitum carbohydrate side with fixed amount of protein: Ad libitum macaroni pasta with vegetarian substitute meatballs (25 g protein)
  Interventions: Other: Ad libitum macaroni pasta with vegetarian substitute meatballs

INTERVENTIONS:
Other: Ad libitum full-fat French fries with beef meatballs — Participants will consume 1 of the 6 treatment meals at each of the 6 study sessions in random orders such that by the end of the study, they will have consumed all 6 treatments.
  Participants will be given 30 minutes to consume the treatment meal and will be instructed to eat all the meatballs but to eat the French fries ad libitum (250 g), until comfortably full, simulating "at home" meal consumption. After providing the participants with the first plate of 250 g French fries and about 120 g meatballs (25 g protein), additional plates of freshly cooked French fries (250 g) alone will be provided 10 and 20 min later and they will be given 30 min to complete the treatment meal. Each treatment will be served with water.
  Arms: Ad libitum full-fat French fries with beef meatballs
Other: Ad libitum instant mashed potatoes with beef meatballs — Participants will consume 1 of the 6 treatment meals at each of the 6 study sessions in random orders such that by the end of the study, they will have consumed all 6 treatments.
  Participants will be given 30 minutes to consume the treatment meal and will be instructed to eat all the meatballs but to eat the mashed potatoes ad libitum (250 g), until comfortably full, simulating "at home" meal consumption. After providing the participants with the first plate of 250 g mashed potatoes and about 120 g meatballs (25 g protein), additional plates of freshly cooked mashed potatoes (250 g) alone will be provided 10 and 20 min later and they will be given 30 min to complete the treatment meal. Each treatment will be served with water.
  Arms: Ad libitum instant mashed potatoes with beef meatballs
Other: Ad libitum macaroni pasta with beef meatballs — Participants will consume 1 of the 6 treatment meals at each of the 6 study sessions in random orders such that by the end of the study, they will have consumed all 6 treatments.
  Participants will be given 30 minutes to consume the treatment meal and will be instructed to eat all the meatballs but to eat the macaroni pasta ad libitum (250 g), until comfortably full, simulating "at home" meal consumption. After providing the participants with the first plate of 250 g macaroni pasta and about 120 g meatballs (25 g protein), additional plates of freshly cooked macaroni pasta (250 g) alone will be provided 10 and 20 min later and they will be given 30 min to complete the treatment meal. Each treatment will be served with water.
  Arms: Ad libitum macaroni pasta with beef meatballs
Other: Ad libitum full-fat French fries with vegetarian substitute meatballs — Participants will consume 1 of the 6 treatment meals at each of the 6 study sessions in random orders such that by the end of the study, they will have consumed all 6 treatments.
  Participants will be given 30 minutes to consume the treatment meal and will be instructed to eat all the meatballs but to eat the French fries ad libitum (250 g), until comfortably full, simulating "at home" meal consumption. After providing the participants with the first plate of 250 g French fries and about 120 g vegetarian "meatballs" (25 g protein), additional plates of freshly cooked French fries (250 g) alone will be provided 10 and 20 min later and they will be given 30 min to complete the treatment meal. Each treatment will be served with water.
  Arms: Ad libitum full-fat French fries with vegetarian substitute meatballs
Other: Ad libitum instant mashed potatoes with vegetarian substitute meatballs — Participants will consume 1 of the 6 treatment meals at each of the 6 study sessions in random orders such that by the end of the study, they will have consumed all 6 treatments.
  Participants will be given 30 minutes to consume the treatment meal and will be instructed to eat all the meatballs but to eat the mashed potatoes ad libitum (250 g), until comfortably full, simulating "at home" meal consumption. After providing the participants with the first plate of 250 g mashed potatoes and about 120 g vegetarian "meatballs" (25 g protein), additional plates of freshly cooked mashed potatoes (250 g) alone will be provided 10 and 20 min later and they will be given 30 min to complete the treatment meal. Each treatment will be served with water.
  Arms: Ad libitum instant mashed potatoes with vegetarian substitute meatballs
Other: Ad libitum macaroni pasta with vegetarian substitute meatballs — Participants will consume 1 of the 6 treatment meals at each of the 6 study sessions in random orders such that by the end of the study, they will have consumed all 6 treatments.
  Participants will be given 30 minutes to consume the treatment meal and will be instructed to eat all the vegetarian meatballs but to eat the macaroni pasta ad libitum (250 g), until comfortably full, simulating "at home" meal consumption. After providing the participants with the first plate of 250 g macaroni pasta and about 120 g meatballs (25 g protein), additional plates of freshly cooked macaroni pasta (250 g) alone will be provided 10 and 20 min later and they will be given 30 min to complete the treatment meal. Each treatment will be served with water.
  Arms: Ad libitum macaroni pasta with vegetarian substitute meatballs

SUMMARY:
The proposed study aims to simulate a meal eaten at home, where meals will provide a fixed amount of protein from beef or vegetarian substitute "meat" balls with ad libitum access to one of mashed potatoes, full-fat fries, or pasta. Postprandial glycemia (PPG), insulin, active ghrelin, satiety, amino acid response and food intake (FI) at the meal and again 3h later (after an ad libitum pizza meal) will be measured. In addition, post-meal PPG and satiety will be measured for one hour after the second meal.

DETAILED DESCRIPTION:
A total of 30 participants (15 males, 15 females) will be recruited in this study at the University of Toronto. Each participant will attend 6 study sessions where they will consume meals consisting of a fixed amount of beef or vegetarian substitute "meat" balls providing 25 g protein with ad libitum access to one of mashed potatoes, fried French fries, or pasta. Questionnaires will be filled out to assess their recent food intake, physical activity, sleep quality, stress level, appetite, physical comfort, and energy/fatigue level, as well as palatability of the food.

Blood samples will be collected at fasting and at various time points over a 3 hour period after eating the meals to measure blood glucose, insulin, active ghrelin and amino acid concentrations. After 3 hours, participants will receive an ad libitum pizza meal to assess their food intake compensation. Post-meal PPG and satiety will be measured for one hour after the pizza meal.

Study hypothesis:

1. Consumption of potatoes in their most usual forms (mashed or deep fried), when compared with pasta in either meat or vegetarian based meals result in lower FI at the meal and lower PPG and insulin.
2. Compensation for the reduced FI in the mashed potato meal does not occur at a pizza meal 3h later.
3. Lower PPG and insulin post-test meal and second meal will be found.
4. The amino acid profile of different meals will be reflected in post-prandial plasma levels and the amino acid response to vegetarian based meals with potatoes will be more balanced compared to the vegetarian based meals with pasta.

Primary objective:

To investigate the effects of potato consumption served with either meat or vegetarian substitute "meat" on meal-time FI and PPG, insulin, satiety and FI compensation at a later meal in healthy and normal weight adults. FI and PPG are primary outcomes and satiety, insulin, active ghrelin, amino acid response and FI compensation are secondary outcomes.

Specific Objectives:

Objective 1: To simulate at home-style meals and determine their effects on FI, satiety, PPG, and insulin, over three hours. Meals will be served with a fixed amount of beef or vegetarian substitute "meat" balls providing 25 g protein with ad libitum access to one of mashed potatoes, fried French fries, or pasta.

Objective 2: To determine the effect of at home-style meals with beef or a vegetarian substitute with mashed potatoes on FI compensation at an ad libitum pizza meal 3h later. Post-meal PPG and satiety will be measured for one hour.

Objective 3: To compare the amino acid response for 3 h after the meat and vegetarian based meals served with mashed potatoes, French fries, or pasta.

ELIGIBILITY:
Inclusion Criteria:

* > 18 and < 45 years of age
* BMI > 18.5 and < 24.9 kg/m2
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the study.
* Willing to maintain current dietary supplement use throughout the study. On test days, subject agrees not to take any dietary supplements until dismissal from the Nutrition Intervention Center. Failure to comply will result in a rescheduled test visit.
* Willing to abstain from alcohol consumption for 24h prior to all test visits.
* Willing to refrain from marijuana/ edibles use for the duration of the study (approximately 6 weeks).
* Willing to avoid vigorous physical activity for 24h prior to all test visits.
* Understanding the study procedure and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Smoking
* Thyroid problems
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, a malabsorptive syndrome, pancreatitis, gallbladder or biliary disease.
* Presence of a gastrointestinal disorder or surgeries within the past year.
* Known to be pregnant or lactating.
* Unwillingness or inability to comply with the experimental procedures and to follow our safety guidelines.
* Known intolerances, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits (i.e Atkins diet, very high protein diets, etc.) or restrained eaters, identified by a score of ≥ 11 on the Eating Habits Questionnaire
* Uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg) as defined by the average blood pressure measured at screening.
* Weight gain or loss of at least 10lbs in previous three months.
* Excessive alcohol intake (more than 2 drinks per day or more than 9 drinks per week).
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose or that could affect the outcome of the study as per investigator's judgment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Glucose Levels | Starting at the beginning of each session (0 minutes before consumption of treatment meal) and every 15-30 minutes up to 180 - 240 minutes (time of completion of each session).
  Blood glucose level (mmol/L) is measured using finger prick capillary blood samples or intravenous blood samples.
Food Intake | After 30 minutes of the treatment meal start.
  Food intake at the treatment meal time will be measured by weighing the carbohydrates (CHO) sides plates after the assigned meal time.

SECONDARY OUTCOMES:
Change in Insulin Levels | Starting at the beginning of each session (0 minutes before consumption of treatment meal) and every 30 minutes up to 180 - 240 minutes (time of completion of each session).
  Level of blood insulin (μU/mL) is measured using finger prick capillary blood samples or intravenous blood samples.
Change in Active Ghrelin Levels | Starting at the beginning of each session (0 minutes before consumption of treatment meal) and every 30 minutes up to 180 - 240 minutes (time of completion of each session).
  Active ghrelin hormone concentrations (μmol/L) is analyzed in intravenous blood samples.
Change in Amino Acid Response (Protein quality) | Starting at the beginning of each session (0 minutes before consumption of treatment meal) and every 30 minutes up to 180 - 240 minutes (time of completion of each session).
  Amino acid concentrations (μmol/L) is analyzed in intravenous blood samples to determine amino acid release.
Food Intake Compensation | at 180 minutes after the treatment meals.
  The food intake compensation after the second meal (ad libitum pizza meal) will be measured (g).
Change in Subjective Appetite | up to 180 - 240 minutes (time of completion of each session)
  Motivation to Eat Adaptive Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Change in Physical comfort | up to 180 - 240 minutes (time of completion of each session)
  Physical Comfort Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Change in Energy Level | up to 180 - 240 minutes (time of completion of each session)
  Energy Level Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Treatment palatability | Immediately after treatment meal consumption
  Treatment Palatability Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Change in Fatigue Level | up to 180 - 240 minutes (time of completion of each session)
  Fatigue Level Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto - Department of Nutritional Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amr AM, Anderson GH, Vien S, Fabek H. Potatoes Compared with Rice in Meals with either Animal or Plant Protein Reduce Postprandial Glycemia and Increase Satiety in Healthy Adults: A Randomized Crossover Study. J Nutr. 2024 Oct;154(10):2999-3011. doi: 10.1016/j.tjnut.2024.08.017. Epub 2024 Aug 23. PMID 39182847